CLINICAL TRIAL: NCT06884176
Title: Complication Rates Associated With Central Venous Catheters Versus Midline Catheters: A Randomized Control Trial
Brief Title: CVCs Versus Midline Catheters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Jacobi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-16724
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Central Venous Catheter; Midline Catheter; Complication of Catheter
Keywords: midline catheter; central venous catheter; central line related bloodstream infection

STUDY DESIGN:
Intervention Model Description: randomized to one of two therapies, central venous access or midline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- central venous catheter (Active Comparator): If randomized to this group, patients will receive a triple lumen central venous catheter
  Interventions: Device: Ultrasound Guided Central Venous Catheter
- Midline catheter (Active Comparator): If randomized to this group, patients will receive a single lumen midline catheter
  Interventions: Device: Ultrasound Guided Midline Catheter

INTERVENTIONS:
Device: Ultrasound Guided Central Venous Catheter — Patients randomized to this arm will receive an ultrasound guided central venous catheter. The catheter is 20cm in length.
  Arms: central venous catheter
Device: Ultrasound Guided Midline Catheter — Patients randomized to this arm will receive an ultrasound guided midline catheter. The catheter is 8-10cm in length.
  Arms: Midline catheter

SUMMARY:
The goal of this clinical trial is to learn if midline catheters can reduce adverse patient outcomes in adult patients requiring a single vasopressor. The main questions the study aims to answer are:

* Do midline catheters reduce the rates of catheter-related bloodstream infections as compared to central venous catheters?
* Do midline catheters reduce the rates of deep venous thrombosis as compared to central venous catheters? Researchers will compare midline catheters to central venous catheters to see if there is a reduction in these events.

Participants will be randomized to the midline catheter group or the central venous catheter group. The catheters will be part of standard of care for vasopressor therapy. The participants will be followed for 30 days.

DETAILED DESCRIPTION:
Within the United States, around 5 million central venous catheters (CVCs) and 150 million peripheral catheters are inserted annually. A 2015 surveillance survey across 10 U.S. states revealed that 4% of hospitalized patients had 1 or more healthcare-associated infections, with 25.6% reported as device-associated infections. Device-associated infections included catheter-related bloodstream infection (CRBSI), catheter-associated urinary tract infections, and ventilator-associated pneumonia. In addition to increased rates of CRBSI, CVCs are associated with upper extremity deep venous thrombosis (DVT). Peripherally inserted central catheters (PICCs) have previously been proposed as an alternative to CVCs to avoid these complications. However, due to the increasing lumen diameter of PICCs, increased rates of catheter-related thrombosis as compared to CVCs have been reported. In contrast to PICCs where the catheter tip ends at the cavo-atrial junction near the right atrium, midline catheters are peripheral vascular devices inserted into the upper extremity veins that terminate at or below the axillary vein. As midlines terminate prior to the large vasculature of the chest, studies have demonstrated lower rates of CRBSI or DVTs as compared to the reported incidence of such complications with PICCs or CVCs. To date, there have been no large-scale randomized control trials comparing CVC and midline complication rates, including thrombosis, CRBSI, central-line associated readmission, and overall patient mortality.

The authors plan to conduct a parallel, 2-group, open-label randomized control trial at a single urban academic center. A convenience sample of adult patients will be obtained over the course of 1 year. Patients with single vasopressor requirements will be subject to enrollment. Patients will be enrolled in the study by clinicians participating in their care who are involved in the placement of the catheter (midline or CVC). Informed consent will take place in the emergency department (ED) prior to the catheter placement. Clinicians will ask patients who are being treated whether they are interested in the study. Study team members will then approach interested patients to obtain consent for the research.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age being treated in the Emergency Department at Jacobi Medical Center

  * Have an upper extremity (left or right arm) that can accept a midline catheter
  * Able to provide consent (patient or health care proxy)
  * Clinical team believes the patient will require inpatient admission at the time of needing intravenous access
  * Requires a central line or midline catheter as an expected requirement of care
* Patients requiring a single vasopressor due to hypotension

Exclusion Criteria:

* Patients in cardiac arrest (prior to achieving ROSC)
* Patients with infection or burns at both upper extremities
* Patient expected to be discharged from the hospital within 24 hours
* Prisoner
* Pregnancy
* Children less than 18 years of age
* The patient is known or is suspected to be allergic to materials contained in the device
* Patients known to have bacteremia
* Patients with existing central venous catheter
* Patients without the ability to consent (or no health care proxy to consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of catheter related bloodstream infections (CRBSI) within 28 days of placement | Up to 28 days from placement of catheter
  The number of CRBSIs will be determined by clinical signs of infection (i.e., fever, chills, leukocytosis or hypotension) and at least one positive blood culture within 28 days of placement of catheter. The total number of CRBSIs will be recorded per study arm.

SECONDARY OUTCOMES:
Number of catheter failures | Up to 28 days from catheter placement
  Any mechanical failures (accidental withdrawal or dislodgement, breakage, occlusion) will be documented. The total number of mechanical failures will be recorded, 1 or more per patient, by study arm. The type of mechanical failures will not be itemized.
Total number of replacement catheters | Up to 28 days
  The total number of replacement IV catheters required will be documented. This will be assessed based on each study arm (midline and central line).
Total number of upper extremity deep venous thrombosis events | From catheter insertion up to hospital discharge, up to 28 days from catheter insertion.
  This is defined as symptomatic or asymptomatic DVT, verified by ultrasound or computed tomography. The total number of upper extremity DVT events will be recorded by study arm.
Number of catheter leakage events | Up to 28 days from catheter placement
  Catheter leakage events is defined as leakage of blood or fluids from the puncture site. The total number of catheter leakage events will be recorded by study arm.
Number of catheter infiltration events | Up to 28 days from catheter insertion
  Catheter infiltration events is defined as infiltration/swelling or pain around the insertion site with medication or fluid administration. The total number of catheter infiltration events will be recorded by study arm

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Dhillon, MD, Principal Investigator — Jacobi Medical Center, Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 12 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)

REFERENCES:
- [Background] Li X, Zhang H, Li H, Sun W. Comparison of complications and indwelling time in midline catheters versus central venous catheters: A systematic review and meta-analysis. Int J Nurs Pract. 2024 Dec;30(6):e13301. doi: 10.1111/ijn.13301. Epub 2024 Sep 3. PMID 39225710
- [Background] Mushtaq A, Navalkele B, Kaur M, Krishna A, Saleem A, Rana N, Gera S, Chandramohan S, Surapaneni M, Chopra T. Comparison of complications in midlines versus central venous catheters: Are midlines safer than central venous lines? Am J Infect Control. 2018 Jul;46(7):788-792. doi: 10.1016/j.ajic.2018.01.006. Epub 2018 Mar 7. PMID 29525366
- [Background] Urtecho M, Torres Roldan VD, Nayfeh T, Espinoza Suarez NR, Ranganath N, Sampathkumar P, Chopra V, Safdar N, Prokop LJ, O'Horo JC. Comparing Complication Rates of Midline Catheter vs Peripherally Inserted Central Catheter. A Systematic Review and Meta-analysis. Open Forum Infect Dis. 2023 Jan 18;10(2):ofad024. doi: 10.1093/ofid/ofad024. eCollection 2023 Feb. PMID 36751645
- [Background] Swaminathan L, Flanders S, Horowitz J, Zhang Q, O'Malley M, Chopra V. Safety and Outcomes of Midline Catheters vs Peripherally Inserted Central Catheters for Patients With Short-term Indications: A Multicenter Study. JAMA Intern Med. 2022 Jan 1;182(1):50-58. doi: 10.1001/jamainternmed.2021.6844. PMID 34842905
- [Background] Tripathi S, Kumar S, Kaushik S. The Practice and Complications of Midline Catheters: A Systematic Review. Crit Care Med. 2021 Feb 1;49(2):e140-e150. doi: 10.1097/CCM.0000000000004764. PMID 33372744
- [Background] Chopra V, Kaatz S, Swaminathan L, Boldenow T, Snyder A, Burris R, Bernstein SJ, Flanders S. Variation in use and outcomes related to midline catheters: results from a multicentre pilot study. BMJ Qual Saf. 2019 Sep;28(9):714-720. doi: 10.1136/bmjqs-2018-008554. Epub 2019 Mar 18. PMID 30886119
- [Background] Trerotola SO, Stavropoulos SW, Mondschein JI, Patel AA, Fishman N, Fuchs B, Kolansky DM, Kasner S, Pryor J, Chittams J. Triple-lumen peripherally inserted central catheter in patients in the critical care unit: prospective evaluation. Radiology. 2010 Jul;256(1):312-20. doi: 10.1148/radiol.10091860. PMID 20574104
- [Background] Bonizzoli M, Batacchi S, Cianchi G, Zagli G, Lapi F, Tucci V, Martini G, Di Valvasone S, Peris A. Peripherally inserted central venous catheters and central venous catheters related thrombosis in post-critical patients. Intensive Care Med. 2011 Feb;37(2):284-9. doi: 10.1007/s00134-010-2043-x. Epub 2010 Sep 21. PMID 20857280
- [Background] Wall C, Moore J, Thachil J. Catheter-related thrombosis: A practical approach. J Intensive Care Soc. 2016 May;17(2):160-167. doi: 10.1177/1751143715618683. Epub 2015 Dec 3. PMID 28979481
- [Background] Magill SS, Edwards JR, Bamberg W, Beldavs ZG, Dumyati G, Kainer MA, Lynfield R, Maloney M, McAllister-Hollod L, Nadle J, Ray SM, Thompson DL, Wilson LE, Fridkin SK; Emerging Infections Program Healthcare-Associated Infections and Antimicrobial Use Prevalence Survey Team. Multistate point-prevalence survey of health care-associated infections. N Engl J Med. 2014 Mar 27;370(13):1198-208. doi: 10.1056/NEJMoa1306801. PMID 24670166